CLINICAL TRIAL: NCT01845519
Title: Feasibility of a Technology-based Intervention to Reach Inactive Breast Cancer Survivors and Objectively Track Step Activity.
Brief Title: Step by Step: A Tailored Walking Intervention for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leanne Kaye (Other)
Collaborators: UNC Lineberger Comprehensive Cancer Center (Other); University of North Carolina (Other)
Responsible Party: Sponsor-Investigator, Leanne Kaye, Doctoral Candidate, UNC Lineberger Comprehensive Cancer Center
Organization: UNC Lineberger Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 121775
Record Dates: First submitted 2013-04-25; First posted 2013-05-03 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2013-12

CONDITIONS: Sedentary Lifestyle; Breast Neoplasms; Survival Rate (Survivorship)
MeSH Terms: conditions — Sedentary Behavior; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Group (Experimental)
  Interventions: Behavioral: Tailored Email
- Targeted Group (Active Comparator)
  Interventions: Behavioral: Targeted Email

INTERVENTIONS:
Behavioral: Tailored Email — Participants will receive tailored emails.
  Arms: Tailored Group
Behavioral: Targeted Email — Participants will receive targeted emails.
  Arms: Targeted Group

SUMMARY:
This study aims to recruit post-treatment breast cancer survivors for a 12-week 2-arm randomized walking intervention. All intervention materials will be delivered electronically.

The investigators hypothesize that at the end of 12-weeks, participants randomized to the intervention group will engage in more weekly steps than those participants randomized to the comparison group.

DETAILED DESCRIPTION:
More than two-thirds of breast cancer survivors are physically inactive. Inactivity is known to negatively impact both morbidity and mortality, and is especially pronounced among cancer survivors. Self-directed interventions targeting inactivity among breast cancer survivors often report clinically insignificant behavior change. More successful behavior change interventions have suggested that tailoring and, more recently, the fostering of intrinsic motivation, may have improved outcomes. However, no interventions to date have utilized these approaches to increase physical activity among sedentary cancer survivors.

AIM 1: Develop and test intervention (tailored) and comparison group (targeted) messages in a sample of sedentary women to determine message acceptability.

AIM 2: Determine the efficacy of a 12-week tailored intervention to increase the number of weekly steps taken among sedentary post-treatment breast cancer survivors compared to a 12-week, targeted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 40-70 years of age
* History of breast cancer stage I-II
* 2-10 years post-treatment
* Sedentary
* Technology access and skills
* Regular access to personal computer/ broadband internet and email account
* Comfortability using internet, and web-based tools
* US Resident

Exclusion Criteria:

* Concurrent enrollment in another physical activity/ lifestyle/ weight loss intervention program/study
* Current secondary cancer diagnosis/ treatment
* Inability to ambulate
* Refusal to wear personal activity monitor (FitBit Ultra) for the duration of the study
* Engaging in regular moderate to vigorous physical activity

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference in weekly steps between intervention and comparison group at the end of the intervention (week 12). | 12 weeks
  The primary outcome will be measured using weekly step data as measured by a commercially available accelerometer. The primary outcome will be the difference in weekly steps between the intervention and comparison group at the end of the intervention (week 12).

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Kaye, PhD, Principal Investigator — University of North Carolina; Dianne Ward, Ed.D, Study Director — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center/ University of North Carolina, Chapel Hill, North Carolina, United States